CLINICAL TRIAL: NCT00006061
Title: Study of Phosphatidylcholine in a Patient With Methionine Adenosyltransferase Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: UNC Lineberger Comprehensive Cancer Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15077; UNCCH-GCRC-1405
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Methionine Adenosyltransferase Deficiency; Metabolism, Inborn Errors
Keywords: genetic diseases and dysmorphic syndromes; inborn errors of metabolism; methionine adenosyltransferase deficiency; rare disease
MeSH Terms: conditions — Hypermethioninemia; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Rare Diseases | interventions — Phosphatidylcholines

INTERVENTIONS:
Drug: phosphatidylcholine

SUMMARY:
OBJECTIVES: I. Determine whether plasma choline and breast milk choline levels are low at fasting in a patient with methionine adenosyltransferase deficiency, and if the choline levels are low, determine whether choline levels respond to dietary supplementation with phosphatidylcholine.

II. Determine whether this patient has a fatty liver by magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Blood is drawn for liver function tests and measurement of plasma choline levels and breast milk samples are taken for measurement of breast milk choline levels at fasting and at 1 hour after breakfast on day 1. The patient then undergoes magnetic resonance spectroscopy of the liver to assess liver density and choline compound mass. The patient then receives oral phosphatidylcholine supplement, and plasma and breast milk samples are taken at 3 and 6 hours after the dose. Oral phosphatidylcholine supplements continue for 30 days. The above studies are repeated on day 31.

ELIGIBILITY:
* Patient with methionine adenosyltransferase deficiency who is nursing

Ages: 20 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1
Dates: Start 2000-01; Study Completion 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Zeisel, Study Chair — UNC Lineberger Comprehensive Cancer Center